CLINICAL TRIAL: NCT00408174
Title: A Multicenter, Randomized, Double-Blind, Actively-Controlled Trial to Evaluate the Safety and Efficacy of a New Tablet Formulation and Dosing Regimen of Balsalazide Disodium 3.3 g Bid Versus Mesalamine (5-ASA) as Asacol® 0.8 g Tid in Mildly to Moderately Active Ulcerative Colitis
Brief Title: Balsalazide Disodium vs. Mesalamine in Mildly to Moderately Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BZUC3003
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: IBD; UC; Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — balsalazide

INTERVENTIONS:
Drug: Balsalazide disodium

SUMMARY:
To establish the efficacy and safety of a new tablet formulation and dosing regimen of balsalazide disodium dosed twice daily in achieving clinical improvement in subjects with mildly to moderately active ulcerative colitis after 6 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* mildly to moderately active ulcerative colitis.
* disease extends at least 20 cm from the rectum.
* baseline MMDAI score between 6-10, inclusive, and greater than or equal to 2 on the MMDAI bleeding component and endoscopy/sigmoidoscopy component.
* not taking more than 4.8 grams/day of Asacol, greater than or equal to 6.75 grams/day of Colazal,or 2.4 grams/day of mesalamine or equivalent daily dose using any other 5-ASA products at any time during the 14 days preceding the initiation of study medication.
* if of childbearing potential, negative serum pregnancy test.

Exclusion Criteria:

* subject has a significant medical, including psychiatric, condition which in the opinion of the investigator precludes participation in the study.
* subject has a history of allergy or intolerance to aspirin, mesalamine, or other salicylates.
* subject's UC has worsened or failed to improve during chronic (i.e., at least 7) therapy with greater than or equal to 6.6 g/day days of balsalazide disodium within 30 days of screening
* subject has received chronic (i.e., greater than 15 consecutive days) of immunosuppressive therapy (e.g. azathioprine, 6 mercaptopurine) or corticosteroids within 30 days of screening. Intermittent use of oral or rectal immunosuppressive therapy or corticosteroids within 30 days of screening is permitted. Intravenous use of corticosteroids within 30 days of screening is not permitted.
* subject has received intra-rectal aminosalicylates for greater than 2 consecutive days within 7 days of screening.
* subject has had any prior bowel surgery, except appendectomy or cholecystectomy.
* subject has participated in an investigational drug or device study within the 30 days prior to study.
* subject is pregnant or at risk of pregnancy, or is lactating (female subjects only).
* subject shows evidence of current excessive alcohol consumption or drug dependence.
* subject has a history of human immunodeficiency virus (HIV). Subjects with history of hepatitis B and C will be eligible provided the screening LFTs are within normal limits.
* subject has other infectious, ischemic, or immunologic diseases with GI involvement.
* subject has twice the upper limit of normal (ULN) for any of the following LFTs: alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT), alkaline phosphatase, or total bilirubin (except isolated elevation of unconjugated bilirubin).
* subject has uncontrolled, clinically significant renal disease manifested by 1.5 × ULN of serum creatinine.
* subject has calculated creatinine clearance level of less than or equal to 60 mL/min.
* subject has unstable cardiovascular, coagulopathy or pulmonary disease characterized by a worsening in the disease condition that required a change in treatment or medical care within one (1) month of randomization.
* subject has active malignancy within the last 5 years, except basal cell carcinoma of the skin, or if female, in situ cervical carcinoma that has been surgically excised.
* subject has any condition or circumstance that would, in the opinion of the investigator, prevent completion of the study or interfere with analysis of study results, including history of noncompliance with treatments or visits.
* subject has sclerosing cholangitis.
* subject has positive stool culture for ovum and parasites (O&P) or C. difficile.
* subject has been treated with infliximab, cyclosporine, natalizumab, or methotrexate for ulcerative colitis within the last 30 days prior to screening.
* regular use of NSAIDS except cardioprotective ASA (i.e., less than or equal to 162 mg ASA per day).
* subject has received cell-depleting therapies such as the Adacolumn.
* subject requires antidiarrheal therapy during screening.
* subject has clinical or radiographic findings suggestive of serious UC complications such as toxic megacolon or colonic perforation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of subjects that achieve clinical improvement and improvement in the rectal bleeding subscale of the MMDAI at the end of six weeks of therapy.

CONTACTS AND LOCATIONS:
Locations (88):
- United States (88):
  - Premiere Pharmaceutical Research, Tempe, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Medical Services of Northwest Arkansas, Fayetteville, Arkansas
  - Gastroenterology Associates, Little Rock, Arkansas
  - AGMG Clinical Research Institute, Anaheim, California
  - West Gastroenterology Medical Group, Los Angeles, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Arapahoe Gastroenterology, PC, Littleton, Colorado
  - South Denver Gastroenterology, Lone Tree, Colorado
  - Phoenix Internal Medical Associates, Waterbury, Connecticut
  - Clinical Trials Management of Bocal Raton, Boca Raton, Florida
  - Research Consultants Group, Hialeah, Florida
  - Horizon Institute for Clinical Researcg, Hollywood, Florida
  - Mark Lamet, M.D., Hollywood, Florida
  - Borland-Grover Clinic, Jacksonville, Florida
  - A+ Research, Miami, Florida
  - West Wind'r Research & Development, Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - The Atlanta Center for Gastroenterology, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Atlanta Academic Research, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Digestive Research Associates, Newnan, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Clinical Trials Management, Metairie, Louisiana
  - Digestive Disorders Association, Annapolis, Maryland
  - Maryland Clinical Trials, Annapolis, Maryland
  - Alan Rosen, M.D., Baltimore, Maryland
  - Digestive Disease Associates, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - The Center for Clinical Research, Hagerstown, Maryland
  - Charm City Research, Lutherville, Maryland
  - Coastal Research Associates, Braintree, Massachusetts
  - Gastroenterology Associates of Western Michigan, Grand Rapids, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Henry Ford West Bloomfield, West Bloomfield, Michigan
  - Gastrointestinal Associates, Jackson, Mississippi
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - The GI Group of South Jersey, Vineland, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Long Island Clinical, Great Neck, New York
  - New York Center for Clinical Research, Lake Success, New York
  - Winthrop University Hospital, Mineola, New York
  - Reseach Associates of NY, New York, New York
  - Simon Lichtiger, M.D., New York, New York
  - Asheville Gastroenterology, Asheville, North Carolina
  - Charlotte Gastroenterology & Hematology, PLLC, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Northwest Piedmont Clinical Research, Elkin, North Carolina
  - Carolina Research Center, Greenville, North Carolina
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Gastroenterology Specialists Inc., Canton, Ohio
  - Digestive Health Network, Cincinnati, Ohio
  - Gastrointestinal & Liver Diseases Consultants, PC, Dayton, Ohio
  - AvamarCenter for Endoscopy, Warren, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - West Hills Gastroenterology, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Guthrie, Sayre, Pennsylvania
  - Charleston Gastroenterology Center, Charleston, South Carolina
  - MUSC Digestive Disease Center, Charleston, South Carolina
  - Clin Search, Chattanooga, Tennessee
  - ACE Research Specialists, Hermitage, Tennessee
  - Gastrointestinal Instititute PLLC, Nashville, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - Houston Digestive Diseases Clinci, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - North Texas Gastroenterology, Lewisville, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Liver and Digestive Disease Specialists, Norfolk, Virginia
  - McGuire VAMC, Richmond, Virginia
  - Discovery Research International, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin